CLINICAL TRIAL: NCT06666036
Title: Leveraging and Strengthening Local Systems to Increase First-time Mothers' Use of Postpartum Family Planning and Improve Postnatal Care in Bangladesh: A Cluster Randomized Controlled Trial
Brief Title: Increase First-time Mothers' Use of Postpartum Family Planning in Bangladesh: The Connect Project
Acronym: Connect BD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Save the Children (Other); Save the Children International Bangladesh (Unknown); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NCR203091
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Contraceptive Usage
Keywords: postpartum family planning; first time mothers; modern contraception
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connect Community Level Enhancements (Experimental): At the community level, Connect enhancements build on standard community health worker (CHW) home visits implemented by the government and pre-existing courtyard meetings implemented by the Government of Bangladesh.
  Courtyard meetings are led by CHWs and convened monthly for new mothers and their families. CHWs sensitize participants to postpartum family planning (PPFP) and share the importance of available services from facilities. Connect reinforces the regularity of these meetings. CHWs receive additional training to be sensitized to the needs of first time parents and engage first-time mothers to attend.
  Home Visits: CHWs conduct home visits to women who are pregnant or recently gave birth in their catchment areas. During these visits CHWs provide basic care, information on ANC, PNC and PPFP, and provide access to FP methods. Connect targets home visits to first time mothers and those who gave birth at home. They provide print materials to support PPFP and PNC care.
  Interventions: Behavioral: Connect
- Control (No Intervention): No additional Connect intervention. Pre-existing institutionalized services for expecting and new mothers.

INTERVENTIONS:
Behavioral: Connect — Community level enhancements
  Arms: Connect Community Level Enhancements

SUMMARY:
While a growing body of programs have shown promise to increase uptake of contraception among FTMs, difficulties remain in scaling beyond small pilot areas and institutionalizing within existing systems. Despite the importance of PNC it remains a neglected area within the maternal and newborn health continuum of care in many areas around the world. Programs working to improve coverage of PNC and PNHVs have faced difficulties with insufficient human resources and health systems, suggesting a need for prioritization of care in settings with limited human resources. Connect's approach aims to strengthen existing government health systems and community-level health efforts, including those supported through local and international non-governmental organizations, by developing and testing light-touch "enhancements" with the goal of increasing PPFP and PNC uptake among FTMs. The investigators will evaluate Connect's approach through a cluster randomized control trial.

DETAILED DESCRIPTION:
While a growing body of programs have shown promise to increase uptake of contraception among FTMs, difficulties remain in scaling beyond small pilot areas and institutionalizing within existing systems. Despite the importance of PNC it remains a neglected area within the maternal and newborn health continuum of care in many areas around the world. Programs working to improve coverage of PNC and PNHVs have faced difficulties with insufficient human resources and health systems, suggesting a need for prioritization of care in settings with limited human resources. Connect's approach aims to strengthen existing government health systems and community-level health efforts, including those supported through local and international non-governmental organizations, by developing and testing light-touch "enhancements" with the goal of increasing PPFP and PNC uptake among FTMs. The investigators will evaluate Connect's approach through a cluster randomized control trial.

The overall goal of this study is to add to the evidence base on scalable and efficacious approaches for increasing PPFP adoption and improving timing and uptake of PNC among adolescent and young FTMs in order to increase spacing before subsequent births and improve maternal and neonatal outcomes.

Specifically, this protocol outlines the parameters for the evaluation of the impact of Connect's package of community-level interventions-or "enhancements"-on adoption and continued use of modern PPFP methods and uptake of PNC among adolescent (ages 15-19 years) and young (ages 20-24 years) FTMs. These interventions are enhanced home visits by family welfare assistants (FWA) and FWA-led enhanced courtyard meetings.

FWA enhanced home visits are targeted based on identification of at-risk mother-baby dyads through a risk-stratification algorithm to ensure home visits to all FTMs who give birth at home and to at-risk mothers, including first time mothers. FWAs performing the enhanced home visits have undergone additional training emphasizing the importance of referring mothers to facility-based providers, encouraging facility delivery, encouraging attendance of courtyard meetings, involving other family members during the visit, and on the specific needs of first-time parents. Invitation cards to go to the nearest facility and mother-baby booklets within formaiton on ANC, PNC, AND PPFP are also provided.

Enhanced courtyard meetings include standard content provided across all locations but Connect reinforces the regularity of these meetings and the FWAs running them will be more sensitized to first-time parents.

Alongside the wider-scale implementation of these enhancements, Connect will support the Ministry of Health as well as local and international NGOs to sustain the enhancements beyond the donor-funded project.

There are four specific aims for understanding the efficacy for Connect's packages:

1. To estimate the causal impact and cost-effectiveness of Connect's community-level interventions (compared to a control) on the primary outcomes of adoption and continuation of modern PPFP methods and timing and uptake of PNC among FTMs ages 15-24 in Noakhali and Madaripur, Bangladesh.
2. To examine the causal impact of Connect's community-level interventions (compared to a control) on secondary outcomes (specified below) among FTMs ages 15-24 in Noakhali and Madaripur, Bangladesh.
3. To compare the impacts of Connect's community-level interventions on adolescent FTMs (ages 15-19) versus young FTMs (ages 20-24).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or has child under 5 months
* Aged 14-25

Exclusion Criteria:

* Younger than 14 or over 25
* Has more than one child or is pregnant and has a child

Ages: 14 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Self-identifies as a first time mother
Enrollment: 2308 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Adoption of Postpartum Family Planning (PPFP): | 12 months
  1. Indicator for adopted a modern contraceptive method within 12 months after giving birth (among women who have given birth).
  Adoption of a modern contraceptive method in the first year after giving birth, among FTMs who have given birth-modern methods are defined here as male condoms, oral contraceptive pills, injectables, and long-active reversible contraception (LARC) methods (implants and intrauterine device (IUD)).
Currently using PPFP | 12 months
  2. Currently using a modern contraceptive method (among women who have given birth). Modern methods are defined here as male condoms, oral contraceptive pills, injectables, and long-active reversible contraception (LARC) methods (implants and intrauterine device (IUD)).
Postnatal Care uptake | 12 months
  3. Indicator for received any PNC, among FTMs who have given birth. Uptake of facility-based PNC for mother and baby. Care that is reported to be a PNC visit but occurs outside of a health facility is not considered a PNC visit for these indicators.
Timing of Postnatal Care (PNC) | 12 months
  4. FTM received PNC within 72 hours of delivery, among FTMs who have given birth more than 72 hours ago.
  Care that is reported to be a PNC visit but occurs outside of a health facility is not considered a PNC visit for these indicators.

SECONDARY OUTCOMES:
Adopted or Intention to adopt PPFP | 12 months
  Indicator for adopt or intention to adopt modern PPFP with 12 months after birth: Using or planning to use a modern contraceptive method to delay or avoid pregnancy within first year of child's life, among all FTMs who have given birth within the past 12 months. Modern methods included in this indicator are: male condoms, oral contraceptive pills, injectables, implants, IUDs
Quality of additional PNC | 12 months
  We measure quality in two ways: (1) Using an indicator for quality of any of an FTM's PNC contact that occurred more than 24 hours after delivery, among FTMs who received a PNC contact. The indicator is equal to one if received all 17 content areas measured; (2) using a scale (0-17) of the total number of content areas covered out of 17 during any PNC contact that the FTM received more than 24 hours after birth. this score will be calculated by generating an indicator for each content area equal to one if the content was covered and summing the indicators.
Quality of early PNC | 12 months
  This will be measured in two ways:
  1. Indicator for quality of early PNC contact (within 24 hours of delivery) for FTM, among FTMs who received an early PNC contact
  2. Scale (0-10) indicating the total number of content areas covered out of 10 during an early PNC contact, among FTMs who received an early PNC contact. This score is calculated by generating an indicator for each content area equal to one if it was covered, sum the indicators to generate the overall scale.
Contraceptive Preferences | 12 months
  Contraceptive preferences for modern methods, among all FTMs, measured with an indicator equal to one if the FTM names a modern method (male condom, pill, injectable, implant, IUD) as preferred family planning method if there were no constraints (e.g., cost, access, opinions of others, etc.).
Quality of Family Planning Counselling | 12 months
  Quality score (0-100), among all FTMs who received family planning counseling. A 22-item quality of care index, adapted from Jain et al. (2019) is combined into a weighted additive index where each of 4 domains have equal weight (1) respectful care, (2) method selection, (3) effective use of method selected, and (4) continuity of contraceptive use and care. For each domain, we will construct an indicator equal to one of the care is of "high quality", defined as having a score that is greater than the mean score plus half of the standard deviation
Communication and agency | 12 months
  Indicator for FTM discussed FP with husband/partner or other family member, among all FTMs
PPFP knowledge | 12 months
  PPFP knowledge index of six true/false statements, standardized to the mean and standard deviation of the control group, among all FTMs. The raw index will be the sum of the responses to each individual true/false statement. Raw scores range from 0 to 6, with 6 indicating that all questions were answered correctly. A set of 5 true/false questions adapted from MOMENTUM asked in a random order.
PPFP Attitudes | 12 months
  PPFP attitudes index of eight attitudes, standardized to the mean and standard deviation of the control group, among all FTMs. The raw index will be the sum of the responses to each individual attitude (score ranging from 1 to 5), with a possible maximum score of 40. Higher scores will indicate less restrictive attitudes with regard to family planning.
PNC attitudes | 12 months
  PNC attitudes index of four attitudes, standardized to the mean and standard deviation of the control group, among all FTMs. The raw index will be the sum of the responses to each individual attitude (score ranging from 1 to 5), with a possible maximum score of 20. Higher scores will indicate less restrictive attitudes with regard to PNC.

CONTACTS AND LOCATIONS:
Locations (1):
- Technical Assistance Inc, Cox’s Bāzār, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made publicly available
Supporting Information: Study Protocol, SAP
Time Frame: 2025